CLINICAL TRIAL: NCT01130571
Title: Establishment and Characterization of Patient-Derived Non-Small Cell Lung Cancer Xenografts and Cell Cultures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: NS03/05/09
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Transplantation, Heterologous; Cell Culture Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Non-Small Cell Lung Cancer
  Interventions: Procedure: Xenografts and cell cultures

INTERVENTIONS:
Procedure: Xenografts and cell cultures

SUMMARY:
Xenografts and cell cultures provide sufficient material for analyses at the protein, RNA and DNA level. Patient derived NSCLC xenografts and cell lines are available but none however are Asian in origin. Given the emerging evidence to suggest inter-ethnic differences in NSCLC biology, new models of preclinical drug evaluation should be designed and validated using Asian tumors. Furthermore, such models will allow studies of biological mechanisms of sensitivity and/or resistance and also the study of dynamic regulations under standardized conditions in the Asian context.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 years and above.
* Undergoing a surgical resection of tumor as part of clinical management

Exclusion Criteria:

* Patient or legally acceptable representative unable to provide consent patient in the judgement of the study investigator, is medically unsuitable for this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators for this protocol are clinicians and scientists in the departments of Cardiac/Thoracic and Vascular Surgery, Haematology and Oncology, Pathology, Radiation Oncology, Respiratory Medicine and the Cancer Sciences Institute of Singapore (CSIS) from NUH and NUS with major roles in their departments in the clinical management and/or research of lung cancer. Each will be providing access to clinical information and assisting in the collection and processing of samples, according to their resources and expertise.
Sampling Method: Probability Sample
Dates: Start 2011-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Estimating the world cancer burden: Globocan 2000. Int J Cancer. 2001 Oct 15;94(2):153-6. doi: 10.1002/ijc.1440. No abstract available. PMID 11668491
- [Background] Thun MJ, Hannan LM, Adams-Campbell LL, Boffetta P, Buring JE, Feskanich D, Flanders WD, Jee SH, Katanoda K, Kolonel LN, Lee IM, Marugame T, Palmer JR, Riboli E, Sobue T, Avila-Tang E, Wilkens LR, Samet JM. Lung cancer occurrence in never-smokers: an analysis of 13 cohorts and 22 cancer registry studies. PLoS Med. 2008 Sep 30;5(9):e185. doi: 10.1371/journal.pmed.0050185. Epub 2008 Sep 9. PMID 18788891